CLINICAL TRIAL: NCT01306877
Title: Prospective Single Blinded Randomized Controlled Trial Comparing The Covidien EEA™ Hemorrhoid and Prolapse Stapling Set With DST Series™ Technology Vs. Ethicon PPH03 In A Hemorrhoidopexy Procedure (HEMOSTASIS)
Brief Title: Comparison Study of Surgical Staplers for the Treatment of Hemorrhoids
Acronym: HEMOSTASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVHEPH0109
Record Dates: First submitted 2011-01-28; First posted 2011-03-02 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Hemorrhoids
Keywords: hemorrhoid; hemorrhoid stapler
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EEA Hemorrhoid and Prolapse Stapling Set (Experimental)
  Interventions: Device: EEA Hemorrhoid and Prolapse Stapling Set
- Endosurgery Proximate PPH03 Stapling Set (Active Comparator)
  Interventions: Device: Endosurgery Proximate PPH03 Stapling Set

INTERVENTIONS:
Device: EEA Hemorrhoid and Prolapse Stapling Set — Surgical device
  Arms: EEA Hemorrhoid and Prolapse Stapling Set
Device: Endosurgery Proximate PPH03 Stapling Set — Surgical device
  Arms: Endosurgery Proximate PPH03 Stapling Set

SUMMARY:
The purpose of this study is to demonstrate that the Covidien EEA™ Hemorrhoid and Prolapse Stapling Set for the treatment of hemorrhoids is non-inferior to the competitor device based on the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able to understand and sign Informed Consent Form
* The subject is between 18-85 years of age.
* The subject has (symptomatic) Grade 2-3 Hemorrhoids and is eligible for stapled hemorrhoidopexy

Exclusion Criteria:

* The procedure is needed as revision hemorrhoid surgery.
* Any female patient, who is pregnant, suspected pregnant, or nursing.
* The participant has an active or a history of infection requiring antibiotics at the intended operative site within thirty (30) days prior to the planned surgery date.
* The participant is unable or unwilling to comply with the study requirements, follow-up schedule.
* The participant has a 1 year history of drug or alcohol abuse.
* The participant has a history of venous thrombosis or pulmonary embolism.
* The participant has a history of coagulopathy.
* The participant has taken aspirin, anti-coagulation and/or anti platelet therapies (e.g. Warfarin, Lovenox) within 7 days prior to the planned date of surgery.
* The participant has a history of fecal incontinence
* The participant has had injection therapy, infrared laser treatment or rubber band ligation for treatment of hemorrhoids within 1 month of screening
* The participant has co-morbidities which, in the opinion of the investigator, will not be appropriate for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Marcet, MD, Principal Investigator — University of South Florida
Locations (1):
- USF Tampa General Hospital Dept of Surgery, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EEA Hemorrhoid and Prolapse Stapling Set: EEA Hemorrhoid and Prolapse Stapling Set : Surgical device
- Endosurgery Proximate PPH03 Stapling Set: Endosurgery Proximate PPH03 Stapling Set : Surgical device
Period: Overall Study
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Started | 78 | 71
Completed | 75 | 67
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set | Total
Number analyzed (Participants) | 78 | 71 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (13.8) | 52.1 (13.4) | 53.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 27 | 66
  Male | 39 | 44 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 7 | 12
  White | 66 | 58 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Hemorrhoid Grade [Number; unit: participants] — Hemorrhoid grading is based on the scale from The American Society of Colon and Rectal Surgeons classification where grade IV represents the worst onset of hemorrhoids and grade I is the best case. Surgeons use the following classification to grade subjects in the study. Grades increase in severity with Grade I being better than Grade IV Grade Physical Findings I Prominent hemorrhoidal vessels, no prolapse
  II Prolapse with Valsalva and spontaneous reduction
  III Prolapse with Valsalva requires manual reduction
  IV Chronically prolapsed manual reduction ineffective
  participants
    Grade 1 | 0 | 0 | 0
    Grade 2 | 28 | 20 | 48
    Grade 3 | 50 | 51 | 101
    Grade 4 | 0 | 0 | 0
Smoking History [Number; unit: participants]
  Non-Smoker | 49 | 38 | 87
  Past Smoker | 12 | 24 | 36
  Current Smoker | 17 | 9 | 26
Prior Hemorrhoid Treatment [Number; unit: participants]
  At least 1 Treatment | 29 | 36 | 65
  No Treatment | 49 | 35 | 84
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.94 (17.61) | 27.11 (4.85) | 27.54 (4.97)
Weight [Mean (Standard Deviation); unit: Kg] | 81.69 (17.61) | 81.29 (18.65) | 81.50 (18.05)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Bleeding
Description: Number of subjects who require intervention to stop intraoperative bleeding The analysis is based on the per protocol analysis set. Subjects who were misrandomized for excluded from this analysis therefore, the population here will differ from the participant flow.
Time Frame: Day 0 - time of surgery
Measure: Number; unit: participants
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 76 | 68
participants | 32 | 50
Statistical Analysis 1: Comparison: EEA Hemorrhoid and Prolapse Stapling Set vs Endosurgery Proximate PPH03 Stapling Set; Test type: Non-Inferiority or Equivalence — The objective is to reject H0 at the 0.05 significance level. A one-sided 95% confidence upper limit for PC - PE will be constructed by Newcombe's generalized Wilson score method (Newcombe 1998). H0 will be rejected at the 0.05 significance level if this upper limit is <7%; p = 0.0001, Chi-squared — P-value calculated from per protocol analysis set; Risk Difference (RD) = -0.314, 95% CI 1-sided [upper limit -0.18]

2. Secondary Outcome: Post Operative Pain - (PI-NIRS)
Description: Post-operative pain as change from baseline pain score as measured by an 11-point Pain Intensity Numeric Rating Scale (PI-NRS). The range of the scale is 0-10 with 0 representing no pain and 10 representing the worst possible pain.
  The data represented is the change in baseline score at the different timepoints.
Time Frame: Day 0 minus 60 (baseline), Day 0 (discharge), Day 0 plus 7, Day 0 plus 30, Day 0 plus 90, Day 0 plus 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 78 | 71
units on a scale
  (Day 0 minus 60) Baseline | 2.0 (2.3) | 2.1 (2.6)
  (Day 0) Discharge | 1.0 (2.8) | 0.8 (3.1)
  (Day 0 plus 7) Week 1 | 0.5 (3.1) | 0.3 (3.2)
  (Day 0 plus 30) Month 1 | -1.0 (2.5) | -1.4 (2.8)
  (Day 0 plus 90) Month 3 | -1.5 (2.2) | -1.8 (2.8)
  (Day 0 plus 180) Month 6 | -1.5 (2.3) | -2.0 (2.6)

3. Secondary Outcome: Post-Operative Pain (Analgesic Intake)
Description: post operative pain measured in pos-surgical consumption of strong opioids by the number of participants in the study. Participants are included if they consumed analgesics or strong opiod at anytime during the study.
Time Frame: Day 0, 1 week, 2 week, 1 month, 3 month, 6 month
Measure: Number; unit: participants
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 78 | 71
participants
  Surgery - discharge | 37 | 25
  Discharge - 1 week post op | 29 | 18
  1 week - 2 week post op | 14 | 15
  2 week - 1 month post op | 5 | 2
  1 month - 3 month post op | 2 | 2
  3 month - 6 month post op | 2 | 2

4. Secondary Outcome: Overall Quality of Life - General Health Score
Description: Quality of life was measured by SF-12 questionnaire in change from baseline; the socring range is 0 - 100 with 0 = poor overall health and 100 = excellent overall health
Time Frame: Day 0 minus 60, 1 week, 1 month, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 70 | 62
units on a scale
  baseline | 53.89 (8.31) | 54.58 (8.65)
  1 week | -0.26 (6.27) | -2.13 (5.90)
  1 month | 0.44 (8.06) | -1.05 (6.62)
  3 month | 0.88 (8.46) | -0.05 (6.91)
  6 month | 1.36 (7.93) | -0.72 (6.46)

5. Secondary Outcome: Location of the Staple Line
Description: Distance of staple line to dentate line as measure by surgical ruler
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 78 | 71
mm | 25.94 (8.23) | 24.00 (8.39)
Statistical Analysis 1: Comparison: EEA Hemorrhoid and Prolapse Stapling Set vs Endosurgery Proximate PPH03 Stapling Set; Test type: Superiority or Other; p = 0.1844, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Length of Stay
Description: Length of hospital stay is defined as time of anoscope insertion until discharge
Time Frame: Day 0 time of discharge minus time of admission
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 78 | 71
Hours | 4.16 (6.17) | 4.37 (6.64)
Statistical Analysis 1: Comparison: EEA Hemorrhoid and Prolapse Stapling Set vs Endosurgery Proximate PPH03 Stapling Set; Test type: Superiority or Other; p = 0.5647, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Operative Room (OR) Time
Description: Time of insertion of anoscope to time of anoscope removal after stapleline evaluation
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Number analyzed (Participants) | 78 | 71
minutes | 25.4 (14.5) | 25.6 (13.2)
Statistical Analysis 1: Comparison: EEA Hemorrhoid and Prolapse Stapling Set vs Endosurgery Proximate PPH03 Stapling Set; Test type: Superiority or Other; p = 0.9062, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Two years - January 2011 to Jan 2013
Description: HEEA N=81 is the total population that was intended to be randomized to the study device using the intent to treat modality. The per protocol population once the misrandomized subjects were excluded is N=78
Arm/Group | EEA Hemorrhoid and Prolapse Stapling Set | Endosurgery Proximate PPH03 Stapling Set
Serious Adverse Events (participants affected / at risk) | 2/81 | 3/68
Other Adverse Events (participants affected / at risk) | 65/81 | 40/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EEA Hemorrhoid and Prolapse Stapling Set (N=81) | Endosurgery Proximate PPH03 Stapling Set (N=68)
Faecoloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EEA Hemorrhoid and Prolapse Stapling Set (N=81) | Endosurgery Proximate PPH03 Stapling Set (N=68)
Anorectal Discomfort (Gastrointestinal disorders) | 7 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 19 (21) | 13 (13)
Operative Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 7 (7)
Suture Insertion (Surgical and medical procedures) | 15 (15) | 17 (17)
Hemorrhage (Vascular disorders) | 0 (0) | 8 (9)
Rectal Hemorrhage (Gastrointestinal disorders) | 14 (17) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No